CLINICAL TRIAL: NCT06709001
Title: CROSS: Colombia's Potential Realized: an Observational Study for Stunting
Brief Title: An Observational Study to Assess Malnutrition Risk
Status: Completed | Type: Observational
Sponsor: Abbott Nutrition (Industry)
Collaborators: Children International (Unknown)
Responsible Party: Sponsor
Other Study IDs: HA70
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Quantitative - Children assessed for Malnutrition Risk: Children living in under-resourced communities
- Qualitative - NGOs, Caregivers, CHWs, and PHPs: Involved in the study as a staff or caregiver or have experience with pediatric malnutrition

SUMMARY:
This is a prospective, observational study for assessing malnutrition risk and its characteristics among children aged 1 to 5 living in under-resourced communities in Colombia. There is also a qualitative component that seeks to gain caregiver, community health worker (CHW), public health professional (PHP), and non-for-profit organization (NGO) insights related to malnutrition risk.

ELIGIBILITY:
Quantitative Inclusion Criteria:

* Children aged 1-5 years
* Children's legal guardian agrees to participate in the study
* Full term pregnancy
* Residence in study area attending Children International (NGO) centers

Quantitative Exclusion Criteria:

* Children who have current medical conditions requiring hospitalization: gastrointestinal tract infections or inflammatory bowel disease; active tuberculosis; acute hepatitis B or C; human immunodeficiency virus OR malignancy; cystic fibrosis; immunodeficiency syndromes, congenital abnormalities of the respiratory tract, such as lung and respiratory cilia; an unsuspected foreign body in the respiratory tract; asthma; and known metabolic disorders, renal impairment, or rheumatic diseases and diabetes,
* Congenital condition
* Children with disabilities such as cerebral palsy, autism spectrum disorder, neurodegenerative disorders
* Children with chronic or acute infections e.g. HIV, malaria
* Children who are taking medications or other agents that could potentially affect body weight, including diuretics, appetite stimulants, steroids, and growth hormones.
* Children already enrolled in a nutrition program/intervention that includes a supplement

Qualitative Inclusion Criteria:

* NGO staff taking part in nutrition screenings
* Caregivers taking part in nutrition screenings as part of this study
* Community health workers (CHW) working with pediatric malnutrition risk
* Public health professionals (PHP) working with pediatric malnutrition risk
* Agrees to participate in focus group/survey

Qualitative Exclusion Criteria:

* Not involved in the implementation of the study
* Not involved in working with pediatric malnutrition risk
* Declines participation in focus group/survey

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Between 2-4 under-resourced communities within Colombia
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Anthropometrics - Height/Length | Baseline, 3 Months and 6 Months
  Measured in cm
Anthropometrics - Mid-Upper Arm Circumference (MUAC) | Baseline, 3 Months and 6 Months
  Measured in mm

SECONDARY OUTCOMES:
Anthropometrics - Weight | Baseline, 3 Months and 6 Months
  Measured in kg
Anthropometrics - Head Circumference | Baseline, 3 Months and 6 Months
  Measured in cm
Nutrient Intake | Baseline and 6 Months
  Caregiver completed 24-hour dietary recall
Pediatric Quality of Life Inventory | Baseline and 6 Months
  A 23-item questionnaire rated 0 to 4 where higher scores indicate better health-related quality of life
World Health Organization Quality of Life Brief Version | Baseline and 6 Months
  a 26-item caregiver completed questionnaire scored 0 to 100 where higher scores indicate higher quality of life
Healthcare Resource Utilization | Baseline and 6 Months
  Caregiver completed questionnaire to obtain illness frequency, severity and related missed school/work days. Higher frequency, severity and missed days associated with greater healthcare utilization.

OTHER OUTCOMES:
Focus Groups with NGOs, Caregivers, CHWs, PHPs | Baseline, 3 Months and 6 Months
  Nutrition program feasibility discussion related to nutrition screening and program participation
Staff Insights Questionnaire | 6 Months
  A non-statistical 6-item questionnaire completed by the NGO Staff to obtain feedback on their experience with nutrition screening
Process Outcomes | Baseline, 3 Months and 6 Months
  Enrollment and adherence to nutrition program

CONTACTS AND LOCATIONS:
Overall Officials: Amy Sharn, MS, RDN, LD, Study Chair — Abbott
Locations (1):
- Children International, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No